CLINICAL TRIAL: NCT00731224
Title: A 24-week, Multi-center, Open-label Evaluation of Compliance and Tolerability of the Once-daily 10 cm² Rivastigmine Patch Formulation in Patients With Probable Alzheimer's Disease.
Brief Title: Compliance and Tolerability of Rivastigmine Transdermal Patch 10 cm² in Patients With Probable Alzheimer's Disease.
Acronym: CARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DAU01
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease, rivastigmine, patch
MeSH Terms: conditions — Alzheimer Disease

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rivastigmine transdermal patch

INTERVENTIONS:
Drug: Rivastigmine transdermal patch

SUMMARY:
This study will evaluate compliance, tolerability, safety, efficacy and caregiver burden of rivastigmine patch 10 cm² treatment in people with Alzheimer's disease (MMSE 10-26) initiating therapy for the first time with a cholinesterase inhibitor, and in patients who were unresponsive to previous cholinesterase inhibitor treatment in a community setting.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease according to the NINCDS-ADRDA (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association) and DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) criteria;
* MMSE score of ≥10 and ≤ 26;

Exclusion Criteria:

* Bradycardia (beats per minute less than 50)
* Body weight less than 40 kg;
* Hypersensitivity to cholinesterase inhibitors.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who can reach the target rivastigmine patch size of 10 cm2 and stay on it for at least 8 weeks. | At week 24

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE), Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL), Global Deterioration Scale (GDS), caregiver burden (Zarit Burden Interview). | At baseline, wk 12 and wk 24
Patient compliance (drug accounting) | During 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (36):
- Australia (11):
  - Novartis Investigative Site, East Gosford, New South Wales
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Hornsby, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Chemside, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Ballarat, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Nedlands
- Malaysia (5):
  - Novartis Investigative Site, Johor Bahru, Johor
  - Novartis Investigative Site, Seremban, Negeri Sembilan
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Kuala Lumpur, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Bundang, Seongnam
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (16):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Bursa, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Konya, Turkey
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Atakum / Samsun
  - Novartis Investigative Site, Emek / Ankara
  - Novartis Investigative Site, Etlik / Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Meselik / Eskisehir
  - Novartis Investigative Site, Talas / Kayseri
  - Novartis Investigative Site, Uskudar / Istanbul